CLINICAL TRIAL: NCT04245436
Title: Acute, Double-blind, Adaptively Randomized Treatment With Duloxetine or Escitalopram, Followed by Open-label Naturalistic Follow-up.
Brief Title: Acute and Long-Term Antidepressant Treatment Success in Adolescents With Anxiety (AtLAS-A)
Acronym: AtLAS-A
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Jeffrey Strawn, MD, Associate professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Strawn AtLAS-A
Record Dates: First submitted 2020-01-07; First posted 2020-01-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Anxiety; Depressive Symptoms
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Duloxetine Hydrochloride; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Duloxetine (Active Comparator): Patients randomized to duloxetine, treatment will be initiated at 30 mg qAM through Week 4 (V5) (consistent with the registration trial for duloxetine in pediatric patients with generalized anxiety disorder). Then, duloxetine will be increased to 60 mg qAM at Week 4 (V5) and will be continued at this dose until Week 6 (V6) or the end of the acute phase of the study. Beginning at Week 6 (V6), duloxetine may be increased to 90 mg daily and at Week 8 (V7), may be increased to 120 mg daily.
  Interventions: Drug: Duloxetine
- Escitalopram (Active Comparator): Patients randomized to escitalopram, will initiate treatment at 5 mg qAM for 1 week and then 10 mg qAM (the recommended starting dose for adolescents 12-17 years and the dose used in the pediatric registration trials). After Week 4 (V5), escitalopram will be increased to 15 mg and this dose will be continued until either Week 6 (V6) or the end of the acute phase of the study; however, at Week 6 (V6), escitalopram may be increased to 20 mg qAM based on efficacy.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Duloxetine — Encapsulated duloxetine 30 mg, 60 mg; once-daily
  Other Names: Cymbalta; Irenka
  Arms: Duloxetine
Drug: Escitalopram — Encapsulated escitalopram 5 mg, 10 mg, 15 mg, 20 mg; once-daily
  Other Names: Lexapro
  Arms: Escitalopram

SUMMARY:
Acute, double-blind, adaptively randomized treatment with duloxetine or escitalopram, followed by open-label naturalistic follow-up.

DETAILED DESCRIPTION:
To identify predictors of the magnitude and trajectory of response to flexibly-dosed duloxetine and escitalopram response in adolescents with anxiety, including those with depressive symptoms. And also to examine long-term predictors of sustained response and relapse in adolescents. To examine predictors of developing depressive disorders in anxious adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Written, informed assent and consent.
* Patients, parent/guardian/LAR must be fluent in the English.
* 12 to 17 years of age, inclusive, at Screening.
* Patients must meet DSM-512 criteria for generalized, social and/or separation anxiety disorder and/or panic disorder, confirmed by the MINI-KID.
* Caregiver who is willing to consent to be responsible for safety monitoring of the patient, provide information about the patient's condition, oversee the administration of the investigational product.
* No clinically significant abnormalities on physical examination.
* Negative pregnancy test at Screening in females.
* Negative urine drug screen at Screening.
* Sexually active patients must practice a reliable method of contraception (Section 15.0) that will continue for the duration of the study and for a minimum of 30 days following the end of study participation. Reliable methods of contraception are defined below; other forms of contraceptives (pharmacological and/or non-pharmacological) are not accepted:

  1. Surgical sterilization
  2. Oral contraceptives (e.g. estrogren-progestin combination or progestin)
  3. Transdermally-delivered contraceptives (e.g., Ortho-Evra), depot injections (e.g., Depo-Provera)
  4. Vaginal contraceptive ring (e.g., NuvaRing), contraceptive implants (e.g., Implanon, Norplant II/Jadelle)
  5. An intrauterine device
  6. Diaphragm plus condom.

Exclusion Criteria:

* DSM-512 diagnosis other than generalized anxiety, social anxiety, separation anxiety or panic disorder(s) that is the primary focus of treatment.
* A history of intellectual disability.
* Suicide risk as determined by either: (1) any suicide attempt within the past 6 months and/or (2) significant risk at Visit 1 (Screening) or Visit 2 (Baseline), as judged by the Investigator.
* Allergy, intolerance, non-response or hypersensitivity to escitalopram or duloxetine.
* Subjects taking other medications that require a taper or washout of more than 5 days.
* Patients who have initiated/terminated psychotherapy/behavior therapy within 1 month before Visit 2 (Baseline), or who plan to initiate/change said therapies during the course of the study will be excluded; if the patient is engaged in psychotherapy, it must have been stable for 1 month prior to baseline.
* A clinically-significant medical illness.
* QTc >450 in males / >460 in females (prolonged QTc based on American Heart Association recommendations for Standardization and Interpretation of the EKG81
* Alcohol or substance use disorder within the past 6 months (nicotine use is permitted).
* Positive urine pregnancy test/pregnancy or breast feeding.
* A positive urine drug screen.
* Patients who are unable to swallow capsules.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Pediatric Anxiety Rating Scale (PARS) severity score | Baseline to Week 24 months (Early Term)
  The PARS is a clinician-rated instrument for assessing the severity of anxiety symptoms associated with common anxiety disorders in children and adolescents. The PARS score is derived by summing 5 of the 7 severity/impairment/interference items (2, 3, 5, 6, and 7)
Change from Baseline in the Clinical Global Impression of Severity (CGI-S) | Baseline to Week 10 (Early Term)
  CGI-S is a seven point scale where 1=Normal and 7=Among the most extremely ill patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Strawn, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No